CLINICAL TRIAL: NCT04759105
Title: Autologous Mesenchymal Stem/Stromal Cells for the Treatment of Workers Affected by Chronic Low Back Pain Due to Multilevel InterVErtebral Disc Degeneration: a Phase IIB Randomized Clinical Trial
Brief Title: Efficacy of Intradiscal Injection of Autologous BM-MSC in Worker Patients Affected by Chronic LBP Due to Multilevel IDD
Acronym: ACTIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Center for Outcomes Research and Clinical Epidemiology, Italy (Other)
Responsible Party: Principal Investigator, Gianluca Vadalà, Professor, MD, PhD, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACTIVE trial_(BRIC2018-ID03); 2019-004476-19 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2023-11

CONDITIONS: Intervertebral Disc Degeneration; Chronic Low-back Pain
Keywords: Low back pain; Spine; Intervertebral disc degeneration; Mesenchymal stem cells; Bone marrow
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Therapeutics; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in 2 arms of 26 patients and followed up for 12 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization result will be a treatment code. The treatment code of the patient will be transmitted to local pharmacy. Blinding or masking will be carried out at all stages of packaging and conditioning for shipping following the treatment allocation. Injections used for all groups will be clear and indistinguishable from each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous BM-MSC injection (Experimental): Two interventions:
  * Bone marrow harvesting from the posterior superior iliac crest region
  * Single injections of a dose of 15 million of autologous BM-MSC each disc affected by IDD (up to 4 discs) via imaging control
  Interventions: Drug: Autologous BM-MSC
- Sham Procedure (Sham Comparator): Two sham procedures:
  * Simulated bone marrow harvesting without insertion into the posterior iliac crest region
  * Simulated injection under only local anaesthesia without disc injection, without placebo injection.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: Autologous BM-MSC — intradiscal injection of autologous bone marrow mesenchymal stromal/stem cells
  Other Names: Treated
  Arms: Autologous BM-MSC injection
Other: Sham Procedure — anaesthesia, no disc injection, no placebo injection
  Other Names: Sham
  Arms: Sham Procedure

SUMMARY:
ACTIVE is a phase II B efficacy monocenter, prospective, randomized, controlled double blinded trial, in which intra-discal autologous adult BM-MSC therapy will be compared with sham treated controls.

This trial will evaluate the efficacy of intradiscal injection of autologous BM-MSCs in workers affected by chronic low back pain (LBP) unresponsive to conventional therapy.

The efficacy will be evaluated 12 months after the treatment in terms of pain relief (VAS, Visual Analog Scale), functionality (ODI, Oswestry Disability Index), quality of life (SF36, Short Form - 36) and work ability index (WAI).

DETAILED DESCRIPTION:
Low back pain (LBP) is the main cause of disability in the world, affecting all occupational sectors with different incidence rates. It is estimated that 60 percent of all workers suffer from LBP during their careers, 10 percent of which become chronic (The Lancet. September 2017). Intervertebral disc degeneration (IDD) is widely recognized as a major contributor to LBP, responsible for at least 40 percent of cases. A key characteristic of IDD is loss of matrix integrity and biomechanical functional failure. Today, no therapy can restore intervertebral disc (IVD) function or provide long-term relief from symptomatic IDD. Current therapies are aimed at pain reduction. When these treatments fail, several types of surgery are performed but they are often related to side effects, disturbance of motion and other biomechanical consequences. New strategies concentrate on treating IDD at an early stage. Encouraging results from phase 1 and 2 clinical trials suggest that cell-based regenerative therapies may provide the world first effective therapy for LBP. LBP patients treated with bone marrow mesenchymal stromal/stem cells (BM-MSC) showed rapid and progressive improvement of functional indexes of 65 percent to 78 percent over 1 year after intradiscal administration without side effect. ACTIVE is an ambitious randomized clinical trial aimed at developing a treatment for IDD based on intradiscal injection of autologous BM-MSC to improve the quality of life of workers and the disability of patients with LBP. ACTIVE main aim is to generate efficacy and safety profiles of single injections of 15 million cells/mL of autologous BM-MSC for each disc affected by IDD (up to 4 discs) versus sham procedure. The regenerative potential of BM-MSC treatment will be assessed by Magnetic Resonance Imaging (MRI) technologies on quarterly basis up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Workers (it means subject has worked at least 2 months, even if not continuously, in the last 6 months)
* Age between 18 and 65 years.
* Signed informed consent.
* Symptomatic chronic LBP due to moderate/severe IDD [modified Pfirrmann score 3-5 (Pfirrmann et al., 2001), Griffith score 4-8 (Griffith et al., 2007)] at max. 4 levels of the lumbar spine unresponsive to conservative treatment, physical and medical for at least 6 months. Physical treatment includes physiotherapy. Medical treatments includes AINS, paracetamol, opioids and myorelaxant.
* Annulus fibrosus intact, demonstrated by MRI.
* Pain baseline > 40 mm on VAS (0- 100).
* NSAID washout of at least 2 days before screening.
* Painkillers washout of at least 24 hours before screening.
* For females of childbearing potential, a negative pregnancy test must be documented at Screening.
* Men and women should use effective contraception during treatment and for at least 12 months after BM-MSC discontinuation. The complete list of contraceptive methods is described in the patient information sheet and in the paragraph 6.5. As a precautionary measure, breast-feeding should be discontinued during treatment with BM-MSC and should not be restarted after discontinuation of BM-MSC.

Exclusion Criteria:

* Non-workers (it means that the person has worked less than 2 months, although not continuously, in the last 6 months)
* Congenital or acquired diseases leading to spine deformations that may upset cell application (scoliosis, isthmus lesion, sacralization and hemisacralization, degenerative spondilolisthesis).
* Spinal segmental instability assessed by dynamic X-Ray.
* Symptomatic facet joints syndrome on MRI (facet joints hyperintensity and hypertrophy evaluated at coronal T2 weighted MRI).
* Prior to the screening visit, has received:

  * Oral corticosteroid therapy within the previous 3 months, OR
  * Intramuscular, intravenous or epidural corticosteroid therapy within the previous 3 months
* Presence of a 5th level with symptomatic IDD (modified Pfirrmann score 3-5, Griffith score 4-8) in the lumbar spine.
* Spinal canal stenosis (Schizas score > B).
* History of spinal infection.
* Lumbar disc herniation and sciatica.
* Endplate abnormality such as Schmorl's Nodes.
* Previous discal puncture or previous spine surgery.
* IDD with Modic III changes on MRI images.
* Patients not eligible to the intravertebral disc surgery.
* Patients who have the risk to undergo a surgery in the next 6 months.
* Patients with local infusion device/devices for corticosteroids.
* Obesity with body mass index (BMI in Kg/size in m2) greater than 35 (obesity grade II).
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
* Abnormal blood tests: hepatic (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] >1.5 × upper limit of normal [ULN]), renal, pancreatic or biliary disease, blood coagulation disorders, anemia or platelet count of <100 × 109/L.
* Pregnant or lactating women, or premenopausal women not using an acceptable form of birth control, are ineligible for inclusion. Contraception will be maintained during treatment and until the end of relevant systemic exposure. Additional pregnancy testing will be performed at the end of relevant systemic exposure. The patients will be required to use contraception from initial treatment administration until 24 months after the last dose of study drug.
* In each case of delayed menstrual period (over 1 month between menstruations), confirmation of absence of pregnancy is strongly recommended. The complete list of contraceptive methods is described in the patient information sheet.
* Positive serology for following infection: Syphilis, HIV, Hepatitis B, or C.
* Contraindication to MRI assessed by the investigator.
* Intolerance or allergy to local anaesthesia.
* Any history of Cancer or immunodeficiency disease.
* Previous transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Pain clinical relief | Baseline to month 12
  Pain clinical reduction of at least 40 percent on Visual Analogic Scale (VAS) between baseline and month 12. VAS pain scale ranges from 0 to 100, where 0 represents no pain and 100 represents the worst pain imaginable.
Functional disability index improvement | Baseline to month 12
  Functional disability reduction of 40 percent on Oswestry Disability Index (ODI, also known as the Oswestry Low Back Pain Disability Questionnaire) at month 12 compared with baseline. ODI scale ranges from 0 to 50 and allows evaluation of disability (0 - 20 percent: minimal disability; 20 - 40 percent: moderate disability; 40 - 60 percent: severe disability; 60 - 80 percent: crippled; 80 - 100 percent: bed-bound or exaggerating their symptoms).
Work ability improvement | Baseline to month 12
  Improvement of 10 percent on Work Ability Index (WAI) at month 12 compared to baseline. The WAI is composed of 7 items and is a validated instrument that assesses the individual work ability of an employee. The total WAI score ranges from 7 to 49 and is calculated by summing up the scores of the 7 items.

SECONDARY OUTCOMES:
Measure pain relief of the patient | Baseline, 1, 3 and 6 months
  Assessed by Visual Analogic Scale (VAS). VAS pain scale ranges from 0 to 100: where 0 represents no pain and 100 represents the worst pain imaginable.
Measure functional disability index of the patient | Baseline, 1, 3 and 6 months
  Assessed by ODI (Oswestry Low Back Pain Disability Questionnaire) scale which ranges from 0 to 50 (0 - 20 percent: minimal disability; 20 - 40 percent: moderate disability; 40 - 60 percent: severe disability; 60 - 80 percent: crippled; 80 - 100 percent: bed-bound or exaggerating their symptoms).
Evaluate disability and quality of life evolution of the patient | Baseline, 1, 3, 6 and 12 months
  Assessed by Short Form-36 Health Survey (SF-36) scores which consist of eight 0-100 scaled scores (vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning and mental health) where a lower score corresponds to more disability and a higher score corresponds to less disability.
Disability and quality of life evolution | Baseline, 1, 3, 6 and 12 months
  Assessed by the patient and the physician on: pain intensity in the lumbar spine (1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme); patient's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor); physician's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor).
Assess rescue painkillers medication | Baseline, 1, 3, 6 and 12 months
  Rescue medication use will be recorded throughout the study duration by a diary file.
Structural assessment | Baseline, 1, 3, 6 and 12 months
  Evolution of affected disc(s) by quantitative Magnetic Resonance Imaging (MRI) density measurements with T2 mapping protocol used as an indication of disc fluid and glycosaminoglycans (GAG) content. In addition MRI spectroscopy will provide an assessment of the chemical changes associated with disc degeneration. The "quality" of the patient's lumbar disc will be monitored non invasively using T2 weighted MRI sagittal images and T1spin/echo MRI at the same time points. Lumbar disc grading will be performed in the sagittal T2 weighted images by two experienced physicians independently, who will review each intervertebral disc (from L1-2 to L5-S1) by the modified Pfirrmann criteria.
Evaluation of cost | 12 months
  Comparison of medical and non-medical costs between the two groups of patients. Resource used in each arm will be collected in physical units in the eCRF at the clinical centre as follows:
  * Acute care medical hospitalisations related to IDD
  * Acute care surgical hospitalisations related to IDD
  * Rehabilitation hospitalisations related to IDD
  * Analgesics
  * Work disruption
Incidence of Adverse Events (AE) | Baseline, 1, 3, 6 and 12 months
  Report of Adverse Events (AE). If the study patients do not spontaneously report any AE occurrence since their last visit, they will be interviewed by the investigator filling a study-specific AE checklist for recording of symptoms and complaints.
Assessment of vital signs | Baseline, 1, 3, 6 and 12 months
  During each visit to the study centre, patients will undergo a physical examination with recording of vital signs (temperature, blood pressure, heart rate, height and weight).
Evaluation of blood and urine analysis | Baseline, 1, 3, 6 and 12 months
  During each visit to the study centre, patients will undergo blood sampling for assessment of routine lab tests (Haematology and Biochemistry) and urine analysis (dipstick).
Analysis of chemical biomarkers for tissue degeneration | Baseline, 3, 6 and 12 months
  Assessment of chemical biomarkers for tissue degeneration through MRI spectroscopy. MRI spectroscopy will be used to provide an assessment of the chemical changes associated with disc degeneration (Zuo et al. 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Vadalà, MD, PhD, Principal Investigator — Campus Bio-Medico University of Rome
Locations (1):
- Campus Bio-Medico University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No